CLINICAL TRIAL: NCT02703090
Title: Assessing the Cortical Response to Noxious and Auditory Stimuli Using Near Infrared Spectroscopy in Subjects Under General Anesthesia
Brief Title: Near Infrared Spectroscopy Cortical Response to Noxious and Auditory Stimuli in Subjects Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Barry Kussman, Senior Associate in Cardiac Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IRB-P00021030
Record Dates: First submitted 2016-03-02; First posted 2016-03-09 (Estimated); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Pain
MeSH Terms: conditions — Pain | interventions — Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Normal saline infusion
  Interventions: Drug: Normal saline
- Drug lower dose (Active Comparator): Remifentanil infusion
  Interventions: Drug: Remifentanil
- Drug higher dose (Active Comparator): Remifentanil infusion
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil
  Other Names: Ultiva
  Arms: Drug higher dose; Drug lower dose
Drug: Normal saline
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The primary aim is to utilize near-infrared spectroscopy (NIRS) in patients under general anesthesia to measure changes in brain blood flow in the bilateral somatosensory cortices and the prefrontal cortices in response to noxious stimulation.

DETAILED DESCRIPTION:
Participants:

Patients with a structurally normal heart scheduled to undergo elective electrophysiology study with catheter ablation of an arrhythmia under general anesthesia were recruited. Forty one patients were enrolled from October 2016 to March 2020. Written informed consent was obtained from the participants or their respective parents/guardians before the study and written assent was obtained from children ≥7 years of age. All study procedures were approved by the Institutional Review Board (IRB-P00021030) of Boston Children's Hospital, Boston, Massachusetts and the study registered with clinicaltrials.gov (NCT02703090).

Randomization, Allocation concealment and blinding:

The hospital research pharmacy used a parallel group design, with block randomization to allocate the patients into either high-dose, low-dose or placebo groups. The clinical staff, research personnel and the patients were unaware of the drug allocated to a particular patient (double-blinded). The decision to unblind was made by the principal investigators (B.K and D.B) and performed by the pharmacy after all the data were acquired, preprocessed and were ready for group level statistical analysis.

Power Analysis:

In our pilot study we had useable data from five of the eleven patients enrolled (45%). The signal of interest had a mean value of -3.764x10-7 Moles with a standard deviation of 2.135x10-7 Moles. This resulted in a standardized effect size of 1.763, when using a zero mean for the null case. In order to achieve a 90% power level for this measure, the number of usable data sets is therefore 8 for each group (total of 24 patients). Considering our previous success rate of 45%, approximately 18 patients will need to be enrolled into each group. However, only 41 patients were able to complete the study, as recruitment was discontinued in March 2020 (a year earlier than projected) due to the Coronavirus pandemic in the United States. The decision to unblind was ultimately made by the principal investigators (B.K and D.B).

fNIRS Acquisition: Changes in hemoglobin concentration during the procedure were recorded using a multichannel continuous wave fNIRS system (CW7, Tech En, Massachusetts, USA) at 690 and 830 nm wavelengths and a sampling frequency of 25 Hz. A customized head probe consisting of 9 optical sources, 12 long-separation optical detectors placed at a distance of 3 cm from the source, and 9 short-separation optical detectors placed at a distance of 0.8 cm from the source, was used. Of the total 33 channels (a channel being a source and detector pair), 24 channels recorded cortical hemoglobin concentration changes and 9 channels recorded physiological hemoglobin concentration changes from extra-cerebral tissue.

Cortical regions of interest:

The 24 channels recorded activity from three different cortical regions viz. left lateral prefrontal cortex (left lPFC), medial frontopolar cortex (mFPC), and right somatosensory cortex (S1). Twelve of these 24 channels were subdivided into six regions of interest (ROI) based on their consistent activation/deactivation to acute nociception in previous studies.

Anesthetic and fNIRS Protocol:

The anesthetic technique was standardized for all patients and the hospital research pharmacy used block randomization to allocate the patients into three groups, Group 1: high-dose remifentanil - 0.5 mcg/kg/min (HD), Group 2: low-dose remifentanil - 0.25 mcg/kg/min (LD), and Group 3: placebo - 0.9% NaCL (PL). The syringes were prepared by the hospital pharmacy and this randomized controlled trial was double-blinded. Following premedication with 2 mg IV midazolam, anesthesia was induced with fentanyl (1.5 mcg/kg up to a maximum of 3 mcg/kg) and a standard dose of propofol titrated to effect. Rocuronium was used for neuromuscular blockade for endotracheal intubation and during the procedure. No additional fentanyl was administered after induction of anesthesia. Anesthesia was maintained with sevoflurane (end-tidal concentration 1% to 4%), adjusting the end-tidal concentration to maintain a Bispectral Index (BIS) (Medtronic, Minneapolis, MN) value between 40 to 60. The test drug infusion and fNIRS monitoring was started after induction of anesthesia while the patient was being prepped and continued until just after the last ablation. A qualified member of the research team continuously monitored the fNIRS data quality throughout the procedure and time-stamped each ablation attempt. A research nurse and/or research assistant manually documented the time, duration and mode (radiofrequency (RF) and/or cryoablation) of each ablation attempt. An audio stimulus prompting a motor task was presented as a control to the patient at least 45 minutes after the start of the procedure.

fNIRS Preprocessing: The fNIRS data was preprocessed and analyzed using in-house scripts in MATLAB R2019b platform. The raw fNIRS data of each subject was first converted from intensity measures to optical density measures. Head-motion correction was then performed using a wavelet-based algorithm. To remove physiological (heart rate, respiration) and other confounding noise sources, a third-order bandpass filter at 0.01-0.15 Hz was applied. Using the modified Beer-Lambert law, optical density measures were converted to oxy-, deoxy- and total-hemoglobin concentrations using hmrOD2conc function in the Homer2 toolbox. A linear temporal regression of the resulting concentration of oxygenated hemoglobin (deltaHbO) time series of each channel was regressed using both the nearest short-separation (physiological channel) signal and the global average of all short-separation signals as the nuisance regressor to remove the effect of extra-cerebral tissue on cortical activity. The residuals of the deltaHbO time series from temporal regression were then used to perform a third-order polynomial fit to regress non-linear drifts and linear trends before further analysis.

fNIRS Data Analysis: The primary outcome measure was the changes in HbO concentration to ablation in placebo vs. remifentanil groups. Therefore, the low and high dose remifentanil subgroups were combined and compared to the placebo group. For those regions that were statistically different between placebo and remifentanil, a post-hoc analysis was performed to identify any differences between the two doses. Secondary outcome measures included the changes in HbO concentration to actual or intended movement, in response to the auditory instruction, and/or the auditory stimuli. Combined analysis of the remifentanil subgroups, and sex-based differences were supplemented to the analysis defined in the protocol on an ad-hoc basis.

Cortical Response to Ablation: The fNIRS hemodynamic response to an ablation event was computed using the block-averaging technique whereby the preprocessed deltaHbO time series was averaged across the total number of ablations for each subject. Since the duration of ablation varied between events and between individuals, each block or trial was defined as the 5 seconds before the start of an ablation event and the 20 seconds following the start of ablation for consistency. Each block was then normalized to the 5 seconds of baseline prior to the start of the ablation in a given block. Hemodynamic-based measures quantified from the block-averaged hemodynamic response to ablation stimuli included: (1) Peak deltaHbO (PeakHbO) which was defined as the maximum HbO concentration change from 4 seconds to 15 seconds following stimulus after subtracting the average HbO concentration change during the initial 0-3 seconds of stimulus; PeakHbO for deactivation to stimulus was computed on the absolute hemodynamic response. (2) Minimum deltaHbO (NadirHbO) was defined as the greatest decrease in HbO concentration in the 15 seconds following the start of ablation; (3) Area under the deltaHbO curve (AUC) was defined as the integral of the HbO curve during the 0-15 seconds period following the start of stimulus. The deltaHbO curve was first scaled using the minimum HbO concentration change for that duration i.e., the NadirHbO becomes the 0 baseline for calculation of AUC. Two sample t-tests were performed to compare the activation measures between placebo and drug groups. A statistical threshold of p<0.05, with multiple comparison correction using Benjamini-Hochberg false-discovery rate (FDR) approach at an alpha of 0.05 was employed to minimize Type-I errors. Multiple comparison correction using FDR was applied for comparisons from all three measures (PeakHbO, NadirHbO, AUC) together. Results that survived the FDR-p threshold are reported to be significant at FDR-corrected p<0.05. Results with p values > FDR-p threshold did not survive multiple comparison correction. The FDR-p threshold, and the original p values are both provided for all comparisons. The 95% confidence intervals were generated using false coverage-statement rate that defines the confidence interval coverage corresponding to the FDR-adjusted p-values. A post-hoc analysis using two sample t-test was performed to identify dose-dependent differences between the remifentanil groups (low-dose vs. high-dose).

Sex-related differences in pain response:

Hemodynamic measures of activation (PeakHbO, NadirHbO, and AUC) during ablation was compared between male (n=16) and female (n=16) participants using a two-way Analysis of Covariance (ANOVA) with sex (males, and females), and drug (drug, and PL) as factors. Effect of biological sex was evaluated due to the altered pain sensitivity and treatment outcomes typically found in male vs female patients. Significant effects of sex were obtained using a statistical threshold of p<0.05, and a multiple comparison correction using Benjamini-Hochberg false-discovery rate was applied at alpha of 0.05 to account for Type-I errors.The 95% confidence intervals were also adjusted for effects that were significant at FDR-corrected p<0.05 using method proposed by Benjamini and Yuketeili.

Cortical Response to non-painful stimuli:

The fNIRS hemodynamic response to auditory stimuli instructing individuals to perform a motor imagery task was also computed using the block averaging technique. The task paradigm lasted for a total of 5 minutes and was presented at least once during the procedure in every subject. A single run with five blocks of stimuli was used to calculate hemodynamic response to auditory stimuli during the procedure. A block was defined as the 5 seconds before auditory cue instructing the patient to start the task (lasting a duration of 1 second), and the 29 seconds following the first auditory cue, including the auditory cue to end task at 15 seconds. Hemodynamic-based measures quantified from the block-averaged hemodynamic response were also defined using the peak change in HbO concentration (PeakHbO), Nadir of deltaHbO concentration (NadirHbO), and AUC measures described earlier. A mixed ANOVA was performed to compare the activation measures during the two types of stimulus between placebo and drug groups and their interaction, where "task" is the within-subject factor with two levels (audio and pain/ablation) and "group" is the between-subject factor with two levels (remifentanil and placebo). A statistical threshold of p<0.05 with multiple comparison correction using Benjamini-Hochberg false-discovery rate approach at an alpha of 0.05 was once again employed. Multiple comparison correction using FDR was applied for comparisons from each measure (PeakHbO, NadirHbO, AUC) separately. As noted earlier, the 95% confidence intervals were adjusted for effects that were significant at FDR-corrected p<0.05 using method proposed by Benjamini and Yuketeili.

ELIGIBILITY:
Inclusion Criteria:

* 12-30 years of age
* Structurally normal heart
* Right-handed
* English-speaking

Exclusion Criteria:

* Unable to cooperate or understand the study
* Neurologic disease
* Diabetes mellitus
* Syndrome of greater than minor severity.
* Smoker
* Scalp or hair does not permit sufficient optical light detection
* Unable to keep his/her head still for a period of 200 consecutive seconds

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry D Kussman, MBBCh, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karunakaran KD, Kussman BD, Peng K, Becerra L, Labadie R, Bernier R, Berry D, Green S, Zurakowski D, Alexander ME, Borsook D. Brain-based measures of nociception during general anesthesia with remifentanil: A randomized controlled trial. PLoS Med. 2022 Apr 22;19(4):e1003965. doi: 10.1371/journal.pmed.1003965. eCollection 2022 Apr. PMID 35452458

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 participants were enrolled in the study. 41 participants completed the study. 3 participants were withdrawn from the study prior to any interventions. 32 participants data were analyzed (of the 41 completing the study, 7 participants were excluded due to poor fNIRS signal quality, and 2 participants were excluded because they received only cryoablations).
Groups:
- Placebo: Normal saline infusion (0.9% NaCl)
- Drug Lower Dose: Remifentanil infusion (0.25 mcg/kg/min)
- Drug Higher Dose: Remifentanil infusion (0.5 mcg/ kg/min)
Period: Overall Study
Arm/Group | Placebo | Drug Lower Dose | Drug Higher Dose
Started | 14 | 14 | 13
Completed | 14 | 14 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Drug Lower Dose | Drug Higher Dose | Total
Number analyzed (Participants) | 14 | 14 | 13 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (2.6) | 15.9 (1.7) | 16.1 (2.3) | 15.8 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 6 | 20
  Male | 9 | 5 | 7 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cortical Oxyhemoglobin Concentrations to Ablation
Description: Changes in peak oxyhemoglobin concentration (PeakHbO) to ablation in placebo vs. the remifentanil groups.
Time Frame: 5 seconds before the start of an ablation event and the 20 seconds following the start of ablation
Population: All enrolled subjects with the exclusion of those with inadequate fNIRS signals (n=7) and those receiving cyroablation (n=2).
Measure: Mean (Standard Error); unit: μM
Groups:
- Placebo: Normal saline infusion
  Normal saline
- Drug lower dose; Drug higher dose: Remifentanil infusion
  Remifentanil
Arm/Group | Placebo | Drug lower dose | Drug higher dose
Number analyzed (Participants) | 9 | 12 | 11
μM
  Peak HbO inferior medial frontopolar cortex (Inf.mFPC) | 0.170 (0.032) | 0.057 (0.021) | 0.085 (0.016)
  Peak HbO superior medial frontopolar cortex (Sup.mFPC) | 0.157 (0.030) | 0.072 (0.019) | 0.077 (0.021)
  Peak HbO anterior superior somatosensory cortex (Ant.SS1) | 0.386 (0.082) | 0.350 (0.095) | 0.185 (0.109)
  Peak HbO posterior superior somatosensory cortex (Pos.SS1) | 0.408 (0.124) | 0.212 (0.074) | 0.130 (0.062)
  Peak HbO inferior lateral prefrontal cortex (Inf.lPFC) | 0.099 (0.035) | 0.003 (0.016) | 0.086 (0.037)
  Peak HbO superior lateral prefrontal cortex (Sup.lPFC) | 0.250 (0.178) | 0.022 (0.028) | 0.156 (0.050)

2. Primary Outcome: Changes in Cortical Oxyhemoglobin Concentrations to Ablation
Description: Changes in nadir oxyhemoglobin concentration (NadirHbO) to ablation in placebo vs. remifentanil groups.
Time Frame: 5 seconds before the start of an ablation event and the 20 seconds following the start of ablation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: μM
Arm/Group | Placebo | Drug lower dose | Drug higher dose
Number analyzed (Participants) | 9 | 12 | 11
μM
  Nadir of deltaHbO Inf.mFPC | -0.141 (0.033) | -0.041 (0.015) | -0.040 (0.017)
  Nadir of deltaHbO Sup.mFPC | -0.130 (0.025) | -0.036 (0.015) | -0.044 (0.020)
  Nadir of deltaHbO Ant.SS1 | -0.292 (0.198) | -0.659 (0.234) | -0.433 (0.147)
  Nadir of deltaHbO Pos.SS1 | -0.585 (0.252) | -0.541 (0.179) | -0.284 (0.076)
  Nadir of deltaHbO Inf.lPFC | -0.105 (0.026) | -0.093 (0.033) | -0.089 (0.031)
  Nadir of deltaHbO Sup.lPFC | -0.237 (0.115) | -0.243 (0.100) | -0.137 (0.048)

3. Primary Outcome: Changes in Cortical Oxyhemoglobin Concentrations to Ablation
Description: Changes in oxyhemoglobin concentration area under the curve (AUC) to ablation in placebo vs. remifentanil groups.
Time Frame: during the 0- to 15-second period following the start of stimulus
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microMolar*seconds
Arm/Group | Placebo | Drug lower dose | Drug higher dose
Number analyzed (Participants) | 9 | 12 | 11
microMolar*seconds
  AUC Inf.mFPC | 25.196 (5.495) | 15.706 (3.909) | 15.634 (3.623)
  AUC Sup.mFPC | 25.399 (5.024) | 15.731 (2.489) | 15.634 (3.623)
  AUC Ant.SS1 | 143.725 (37.211) | 112.650 (24.229) | 95.376 (21.719)
  AUC Pos.SS1 | 155.067 (39.318) | 108.374 (16.526) | 95.199 (24.330)
  AUC Inf.lPFC | 35.787 (8.049) | 35.496 (12.386) | 39.077 (15.493)
  AUC Sup.lPFC | 81.577 (36.490) | 75.484 (30.408) | 41.614 (12.418)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Placebo | Drug Lower Dose | Drug Higher Dose
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02703090/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT02703090/ICF_001.pdf